CLINICAL TRIAL: NCT05785390
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase IIa/IIb Study to Evaluate the Safety, Tolerability, and Efficacy of NP-101 in Treating High-Risk Participants Who Have Tested Positive for Novel Coronavirus 2019.
Brief Title: Study of the Safety, Tolerability and Efficacy of NP-101 in Treating High Risk Participants Who Are Covid-19 Positive.
Acronym: BOSS-002
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The interim analysis results met protocol and SAP predetermined criteria for stopping early due to futility or efficacy.
Sponsor: Novatek Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOSS-Covid-19-002
Record Dates: First submitted 2023-03-23; First posted 2023-03-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: COVID-19
Keywords: COVID-19; High Risk; Outpatient
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase IIb will be a 2 parallel arms, double - blind, randomized, placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Participant, Investigator will all be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Drug Treatment (Experimental): Phase IIa - Dose escalation. 3g cohort and 4.8g cohort run simultaneously, followed by a 6 g cohort. Administered in 600 g capsules of NP-101 for a total daily dose of 3g, 4.8g and 6g adminstered BID. Administered for 14 days.Establish MTDD Phase IIB - Continue study with MTDD as established above.
  Interventions: Drug: NP-101
- Placebo (Placebo Comparator): As above, except dosed with matching placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NP-101 — NP-101 is an organically derived, GMP manufactured product covered under IND #152687.
  Other Names: TQ Formula
  Arms: Active Drug Treatment
Other: Placebo — Identical placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the safety, tolerability, and efficacy of NP-101 in treating high-risk participants who have tested positive for Covid-19. The main question[s] it aims to answer are:

* To evaluate the safety of NP-101, as well as establish the maximum tolerated dose in high risk Covid-19 positive patients.

Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items]. If there is a comparison group: Researchers will compare [insert groups] to see if [insert effects].

DETAILED DESCRIPTION:
This is a Phase IIa/IIb multicenter, interventional, randomized, double-blind, placebo-controlled study designed to evaluate the safety, tolerability, and efficacy of NP-101 in outpatient high-risk COVID-19 positive participants. Blinding roles: Participants, Investigators and Sponsor

The study is comprised of two parts (Phase IIa and Phase IIb) and four cohorts. The first part of the trial (IIa) involves three cohorts and is a dose escalation study designed to select the maximum tolerated dose for use in the second part (IIb) of the study. In the dose escalation (Phase IIa) portion of the trial (n= 60), qualified participants will be enrolled in a parallel dose escalation design and randomized in a 3:1 [active+best supportive care (BSC):placebo+BSC]ratio to one of three cohorts of 20 participants each (15 active +BSC, 5 placebo + BSC). Cohort 1 (15 participants taking 600 mg capsules for a total daily dose of 3 grams of NP-101 plus BSC and 5 participants taking placebo plus BSC), and Cohort 2 (15 participants taking 600 mg capsules for a total daily dose of 4.8 g of NP-101+ BSC and 5 participants taking placebo plus BSC will run concurrently since acceptable safety data for the 3 g dose was obtained in an earlier phase II study.

Cohort 1 will receive either 3 g Total Daily Dose (TDD) of NP-101 + BSC or Placebo+ BSC, Cohort 2 will receive either 4.8 g TDD of NP-101 +BSC or placebo + BSC) and Cohort 3 (15 participants taking 600 mg capsules for a total daily dose of 6 g of NP-101 + BSC and 5 participants taking placebo plus BSC.) Safety will be evaluated according to the terms of the Statistical Analysis Plan (SAP). In the second portion of the trial (Phase IIb), Participants enrolled in Cohort 4 (n= 248) will be randomized in a ratio of 1:1 (active+BSC : placebo+BSC) and will receive the Maximum Tolerated Daily Dose (MTDD) as determined by the parameters set by the SAP and approved by the pharmacovigilance team.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* A resting SpO2 of >93% on room air.
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged 18 and over, presenting with mild to moderate clinical symptoms of Covid- 19 infection (per FDA guidance - see appendix 3) with symptom onset within 5 days prior to the day of randomization
* Positive COVID-19 infection confirmed by RT-PCR within the last 5 days of the day of randomization
* A score of ≥ 2 (moderate) on a minimum of 1 symptom on the PRO Symptom Survey on the day of randomization
* Ability to take oral medication and be willing to adhere to the dosing regimen (Twice a day - BID for 14 days)
* For females of reproductive potential: negative pregnancy test at screening and use of highly effective contraception method during study participation and for an additional 4 weeks after the end of study drug administration
* For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation and for an additional 4 weeks after the end of study drug administration
* Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration
* To be considered high risk, participants should have at least one of the following conditions:

  * age ≥60 years;
  * active cancer
  * chronic kidney disease;
  * chronic lung disease including COPD
  * Obesity (BMI ≥30)
  * serious heart conditions [heart failure, coronary artery disease, or cardiomyopathies];
  * Diabetes (type 1 or type 2)
  * Immunocompromised state (weakened immune system or autoimmune diseases)
  * Chronic liver disease
  * Cystic fibrosis
  * HIV infection
  * Smoking, current or former
  * Sickle cell disease or thalassemia
  * Solid organ or blood stem cell transplant
  * Stroke or cerebrovascular disease

Exclusion Criteria:

* Current or recent (within 4 weeks) treatment with any corticosteroids; however, inhaled steroids, which are used to treat acute or chronic bronchial inflammation, will be permitted
* Severe Covid-19 symptoms (severe per FDA classification - see appendix 3)
* Requires immediate admission to hospital for any reason
* Pregnancy or lactation
* Known allergic reactions to components of black seed oil or thymoquinone
* Treatment with another investigational drug or other investigational intervention within 2 weeks of study start and throughout study duration.
* Significant hepatic disease (ALT/AST> 4 times the ULN); any laboratory parameter >/= 4 times the ULN or platelet count <100,000/µ L or neutrophilic granulocyte absolute count

  o <500/mm3
* History of moderate to severe CKD, (i.e. on hemodialysis or has an estimated glomerular filtration rate less than 45mL/min) at the time of enrollment
* Participants with inflammatory bowel disease (such as Crohn's) that could affect the intestinal absorption of NP-101 enteric coated capsules.
* Known uncontrolled HIV (with a recent viral load > 50 copies/mL or CD4<200 cells/mm3 or known active uncontrolled Hepatitis B (defined as HBsAg-positive or detectable HBV DNA viral load) or known active Hepatitis C (defined as detectable HCV RNA viral load) infection
* Influenza diagnosis (confirmed by testing) during screening or within prior 14 days
* Any uncontrolled condition(s) or diagnosis, both physical or psychological, or physical exam finding that precludes participation, as per investigator
* Current treatment with CYP2C9 substrates (see Appendix 5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Establishment of MTDD | Fourteen days per dose (Phase IIA Only)
  Number of DLTS (Dose Limiting Toxicities) in the NP-101 arm at each dose compared to placebo and the safety threshold
Safety and Tolerability of NP-101 vs Placebo (Phase IIa and IIb) | Through Day 45
  Evaluation of the number of overall adverse events, related adverse reactions, adverse events leading to d/c of study drug and hospitalizations or death.
Time to Sustained Clinical Recovery | Through Day 5
  Measurement of the difference of SCR rates on Day 5 in patients taking the MTDD of NP-101 vs Placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kaseb, MD, Study Director — Novatek Pharmaceuticals
Locations (4):
- United States (4):
  - L&A Morales Healthcare/ Enrique Villa, MD Principal Investigator, Miami, Florida
  - Research Network America, Berwyn, Illinois
  - Clinical Trial Network, Houston, Texas
  - Pearland Family Wellness Clinic, Pearland, Texas

IPD SHARING:
Plan to Share IPD: No